CLINICAL TRIAL: NCT01832727
Title: Phase 1b/2, Multicenter, Open-label Study of Oprozomib and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment halted during phase 2 to reformulate the investigational product
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-001; 20130408 (Other: Amgen); 2013-001169-18 (EudraCT Number)
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; oprozomib; OPZ; ONX 0912; Onyx; proteasome inhibitor; oprozomib tablets
MeSH Terms: conditions — Multiple Myeloma | interventions — ONX 0912; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 180 mg 5/14 Schedule (Phase 1b) (Experimental): Oprozomib 180 mg treatment once daily for 5 consecutive days bimonthly (days 1, 2, 3, 4, and 5 of a 14-day cycle) with 20 mg dexamethasone once daily on days 1, 2, 8, and 9 (referred to as the 5/14 schedule). Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 210 mg 5/14 Schedule (Phase 1b) (Experimental): Oprozomib 210 mg treatment once daily for 5 consecutive days bimonthly (days 1, 2, 3, 4, and 5 of a 14-day cycle) with 20 mg dexamethasone once daily on days 1, 2, 8, and 9 (referred to as the 5/14 schedule). Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  This was the first cohort to enroll participants into the 5/14 schedule. The Cohort Safety Review Committee (CSRC) reviewed safety data and made dose adjustments for oprozomib in 30 mg increments for all cohorts.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 150/180 mg 5/14 Schedule (Phase 1b) (Experimental): Oprozomib 150 mg once daily treatment for 5 consecutive days (days 1, 2, 3, 4, and 5 of a 14-day cycle) followed by a step-up in oprozomib once daily dose to 180 mg starting in cycle 2 and moving forward. Dexamethasone 20 mg once daily was administered on days 1, 2, 8, and 9 of each 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 210 mg 2/7 Schedule (Phase 1b) (Experimental): Oprozomib 210 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  This was the first cohort to enroll participants into the 2/7 schedule. The Cohort Safety Review Committee (CSRC) reviewed safety data and made dose adjustments for oprozomib in 30 mg increments for all cohorts.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 240 mg 2/7 Schedule (Phase 1b) (Experimental): Oprozomib 240 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 270 mg 2/7 Schedule (Phase 1b) (Experimental): Oprozomib 270 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 300 mg 2/7 Schedule (Phase 1b) (Experimental): Oprozomib 300 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Cohort 330 mg 2/7 Schedule (Phase 1b) (Experimental): Oprozomib 330 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone
- Phase 2 300 mg 2/7 Schedule (Experimental): The Cohort Safety Review Committee (CSRC) determined this dose as the recommended phase 2 dose (RP2D). Oprozomib 300 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Oprozomib — Oprozomib tablets were supplied containing 60, 90, or 120 mg of oprozomib. Oprozomib extended release tablets were supplied containing 150, 180, 210, 240, or 270 mg of oprozomib. Both formulations were administered in a single dose on dosing days. The tablet formulation required multiple tablets to reach each dose on dosing days.
  Other Names: OPZ; ONX 0912; oprozomib ER
Drug: Dexamethasone — Dexamethasone was administered as 20 mg tablets in strengths of 4 and 6 mg taken orally. If a participant could not tolerate tablets or tablets were unavailable, 20 mg administered intravenously was substituted.

SUMMARY:
The primary objectives are:

Phase 1b:

* To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of oprozomib given orally, once daily, on 2 different schedules.
* To evaluate safety and tolerability

Phase 2:

* To estimate the overall response rate (ORR).
* To evaluate safety and tolerability

DETAILED DESCRIPTION:
The purpose of the Phase 1b portion of the study was to determine the maximum tolerated dose (MTD), the recommended phase 2 dose (RP2D), safety, and pharmacokinetics (PK) of oprozomib administered orally once daily in combination with dexamethasone, in participants with relapsed and/or refractory multiple myeloma, using a 3 + 3 dose-escalation scheme with and without step-up dosing. The MTD was defined as the highest dose level at which fewer than 33% of participants had a dose-limiting toxicity (DLT).

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of multiple myeloma with measureable disease as indicated by 1 or more of the following:

   * a. Serum M-protein ≥ 500 mg/dL
   * b. Urine M-protein ≥ 200 mg/24 hours
   * c. Only for subjects without measurable serum and urine M-protein, serum free light chain: Involved free light chain (FLC) level ≥ 10 mg/dL, provided serum FLC ratio is abnormal
2. Patients requiring therapy who have relapsed and/or are refractory to their last therapy and have been treated with at least 1, but not more than 5, lines of multiple myeloma therapy. Prior therapy must have consisted of at least 1 regimen that included lenalidomide and/or bortezomib. Patients should be considered to be appropriate candidates for a clinical study by their treating physicians. Relapsed patients must have previously achieved ≥ minimal response (MR) on at least 1 line of therapy, as assessed by the treating physician. Refractory patients are allowed, but it is not required that patients be refractory to their last therapy. Primary refractory patients are allowed in the Phase 1b portion of the study only.
3. Males and females ≥ 18 years of age
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
5. Adequate hepatic function, with bilirubin ≤ 1.5 times the upper limit of normal (ULN) in the absence of Gilbert's disease or hemolysis, aspartate aminotransferase (AST) ≤ 3 times ULN, and alanine aminotransferase (ALT) ≤ 3 times ULN
6. Absolute neutrophil count (ANC) ≥ 1000 cells/mcL, hemoglobin ≥ 7.0 g/dL, and platelet count ≥ 30,000 cells/mcL:

   * a. Patients must not have received platelet transfusions for at least 1 week prior to Screening.
   * b. Screening ANC must be independent of granulocyte colony-stimulating factor and granulocyte-macrophage colony-stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for

     ≥ 2 weeks prior to first dose.
   * c. Patients may receive red blood cell (RBC) transfusions or receive supportive care with erythropoietin or darbepoetin in accordance with institutional guidelines.
7. Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute calculated using the formula of Cockcroft and Gault ([140 - Age] * Mass (kg) / [72 * creatinine mg/mL]). Multiply result by 0.85 if female.
8. Uric acid, if elevated, must be corrected to within laboratory normal range before dosing.
9. Patients must sign a written informed consent form in accordance with federal, local, and institutional guidelines.
10. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to receiving the first dose of study drug and agree to use effective methods of contraception during the study and for 3 months following the last dose of study drug. Postmenopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.
11. Prior carfilzomib is not required but is allowed if a patient had at least 2 cycles of carfilzomib alone or in combination with a dose of at least 20/27 mg/m^2, as long as the patient:

    * a. Had at least a partial response to prior carfilzomib therapy
    * b. Was not removed from carfilzomib therapy due to toxicity, unless approved by the medical monitor
    * c. Was not removed from carfilzomib therapy for progressive disease nor experienced progressive disease within 6 months after any prior carfilzomib therapy.

Key Exclusion Criteria:

1. Radiation therapy within 2 weeks prior to first dose; localized radiation therapy within 1 week prior to first dose
2. Immunotherapy/standard myeloma therapy within 2 weeks prior to first dose (except for antibody therapy, where 6 weeks are required, and alkylator therapy, where 3 weeks are required); prior stem cell transplant (SCT) therapy (autologous SCT within the prior 8 weeks; allogeneic SCT within the prior 16 weeks). Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-versus-host disease (GvHD).
3. Plasmapheresis is not permitted at any time during the Screening period or while the subject is receiving study treatment. If a subject has started screening procedures requiring plasmapheresis, or is anticipated to require plasmapheresis during or after the Screening period, this patient will be considered ineligible and should not be enrolled.
4. Glucocorticoid therapy within 14 days prior to enrollment that exceeds a cumulative dose of 160 mg of dexamethasone or equivalent
5. Participation in an investigational therapeutic study within 3 weeks prior to first dose
6. Prior oprozomib exposure
7. Known hypersensitivity/toxicity or intolerance to dexamethasone
8. Major surgery within 3 weeks prior to first dose
9. Congestive heart failure ([CHF] New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to first dose
10. Uncontrolled hypertension or uncontrolled diabetes
11. Active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to first dose
12. Known or suspected human immunodeficiency virus (HIV) infection or patients who are HIV seropositive
13. Active hepatitis A, B, or C infection
14. History of previous clinically significant GI bleed in the last 6 months prior to first dose
15. Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose
16. Other malignancy within the past 3 years, with the exception of adequately treated basal cell carcinoma of the skin, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast, prostate cancer of Gleason Score of 6 or less with stable prostate specific antigen levels, or cancer considered cured by surgical resection
17. Plasma cell leukemia
18. Female patients who are pregnant or nursing
19. Inability to swallow medication, inability or unwillingness to comply with the drug administration requirements, or GI condition that could interfere with the oral absorption or tolerance of treatment
20. Any contraindication to oral hydration (e.g., significant preexisting comorbidity or fluid restriction)
21. Any clinically significant psychiatric or medical condition that in the opinion of the investigator could increase patient risk or interfere with protocol adherence or a patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (10):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Division of Hematology/ Oncology, UNC at Chapel Hill, Chapel Hill, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - CHRU, Hopital Huriez - Department of Hematology, Lille
  - CHU Hotel Dieu - Service d'Hematologie Clinique, Nantes
  - CHU de NANCY - Hopital de BRABOlS, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Hari P, Paba-Prada CE, Voorhees PM, Frye J, Chang YL, Moreau P, Zonder J, Boccia R, Shain KH. Efficacy and safety results from a phase 1b/2, multicenter, open-label study of oprozomib and dexamethasone in patients with relapsed and/or refractory multiple myeloma. Leuk Res. 2019 Aug;83:106172. doi: 10.1016/j.leukres.2019.106172. Epub 2019 Jun 17. PMID 31229804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 centers in the United States and France.
Pre-assignment Details: Eighty-one subjects were screened; sixteen were not enrolled due to entry criteria violations.
Period: Overall Study
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule
Started | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
Not completed — Adverse Event | 4 | 6 | 1 | 0 | 1 | 1 | 2 | 1 | 9
Not completed — Disease progression | 3 | 0 | 2 | 1 | 3 | 3 | 6 | 2 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all subjects who receive at least 1 dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule | Total
Number analyzed (Participants) | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18 | 65
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 5 | 4 | 2 | 1 | 4 | 2 | 4 | 5 | 6 | 33
  65 - <75 years | 2 | 3 | 0 | 2 | 0 | 3 | 3 | 0 | 7 | 20
  >=75 years | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 2 | 1 | 2 | 3 | 2 | 9 | 27
  Male | 6 | 3 | 2 | 2 | 3 | 4 | 5 | 4 | 9 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 7 | 3 | 4 | 2 | 6 | 8 | 5 | 11 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 8
  White | 8 | 7 | 2 | 3 | 2 | 4 | 7 | 4 | 10 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose-Limiting Toxicities (DLT)
Description: Toxicities (graded per the Common Terminology Criteria for Adverse Events v 4.03) were considered DLTs if judged by the investigator to be related to oprozomib and occurred in the first 14 days of treatment, with treatment at the dose to be studied (i.e., Cycle 1 for continuous dosing or Cycle 2 for step-up dosing). A DLT was categorized as nonhematologic or hematologic. Examples include:
  * Any ≥ Grade 3 nonhematologic AE, with exceptions or qualifications such as Grade 3 nausea, vomiting, diarrhea, or constipation were considered a DLT only if lasting for > 7 days despite optimal supportive care
  * Grade 3 fatigue lasting > 14 days
  * Grade 4 neutropenia: absolute neutrophil count (ANC) < 500 cells/mcL lasting ≥ 7 days
  * Febrile neutropenia: Any single temperature ≥ 38.3°C or a sustained temperature of ≥ 38.0°C for over 1 hour with ≥ Grade 3 neutropenia (ANC < 1000 cells/mcL)
  * Grade 3/4 thrombocytopenia
  * Others specified in the protocol
Time Frame: Day 1 to Day 14 (Cycle 1) for continous dosing and Day 15 to Day 28 (Cycle 2) for step-up dosing
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
Participants
  Participants reporting >=1 DLT | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 2 | 1
  Mental status changes | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypertension | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subarachnoid haemorrhage | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Thrombocytopenia | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Upper respiratory tract infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pain in jaw | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) During Phase 1b and 2
Description: AE defined as any untoward medical occurrence in a clinical trial participant. Treatment-emergent adverse events were defined as adverse events that start on or after the first day of study treatment and within 30 days of the last day of study treatment. An adverse event that was present before the first administration of study treatment and subsequently worsens in severity during treatment was also considered to be treatment-emergent.
  Serious AE defined as AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other significant medical hazard. Severity of AEs assessed according to Common Terminology Criteria for Adverse Events (CTCAE, v4.03) based on the general guideline: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening or disabling; Grade 5: Death related to AE.
  IP=investigational product
Time Frame: Day 1 up to Week 282
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
Participants
  >=1 TEAE | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
  Grade >=3 (severe) | 8 | 5 | 2 | 3 | 3 | 5 | 6 | 5 | 16
  Serious AE | 4 | 2 | 2 | 2 | 1 | 1 | 3 | 0 | 9
  Leading to discontinuation of IP | 4 | 6 | 1 | 0 | 1 | 1 | 2 | 1 | 11
  Fatal AE | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Participants With Treatment-Related, Treatment-Emergent Adverse Events (TEAEs) During Phase 1b and 2
Description: AE defined as any untoward medical occurrence in a clinical trial participant. TEAEs were defined as AEs that start on or after the first day of study treatment and within 30 days of the last day of study treatment. An AE that was present before the first administration of study treatment and subsequently worsens in severity during treatment was also considered a TEAE.
  Investigator assessed AEs for relatedness to study drug. Serious AE defined as AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other significant medical hazard. Severity of AEs assessed according to Common Terminology Criteria for Adverse Events (CTCAE, v4.03) based on the general guideline: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening or disabling; Grade 5: Death related to AE.
  IP=investigational product
Time Frame: Day 1 up to Week 282
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
Participants
  >=1 related TEAE | 9 | 7 | 3 | 4 | 4 | 6 | 8 | 6 | 18
  Grade >=3 (severe) | 8 | 5 | 2 | 2 | 2 | 2 | 4 | 3 | 14
  Serious AE | 3 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 3
  Leading to discontinuation of IP | 3 | 6 | 0 | 0 | 1 | 1 | 1 | 1 | 7
  Fatal AE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Best Overall Response in Phase 2 as Assessed by Investigator
Description: Disease response and progression were determined using the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC), except for minimal response (MR) and near complete response (nCR) which was based on the European Group for Blood and Marrow Transplantation (EBMT) criteria. Evaluations reported were assessed by the investigator for participants in Phase 2.
Time Frame: Screening: Day 14 to Day -1; During study: Day 1 up to 13.16 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
Participants
  Stringent Complete Response (sCR) | 0
  Complete Response (CR) | 1
  Near Complete Response (nCR) | 0
  Very Good Partial Response (VGPR) | 2
  Partial Response (PR) | 9
  Minimal Response (MR) | 1
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 1
  Not Evaluable (NE) | 2
  Unknown | 0

5. Primary Outcome: Percentage of Participants Who Achieved an Overall Response As Assessed by Investigator During Phase 2
Description: The overall response rate (ORR) was defined as the percentage of participants with the best overall response of stringent complete response (sCR), complete response (CR), near complete response (nCR), very good partial response (VGPR), and partial response (PR) as defined by the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC) and modified European Group for Blood and Marrow Transplantation (EBMT) criteria.
Time Frame: Screening: Day 14 to Day -1; During study: Day 1 up to 13.16 months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
percentage of participants | 66.7 [41.0 to 86.7]

6. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Time to Maximum Serum Concentration (Tmax) on Cycle 1, Day 1
Description: PK samples obtained on the following schedule:
  Phase 1b Continuous Dosing, Cycles 1 and 2: Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 8 hours post-dose plus pre-dose on Day 2 Phase 1b Step-up Dosing, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2 Phase 2, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2
Time Frame: Day 1
Population: Safety population
Measure: Median (Full Range); unit: hours
Groups:
- 180 mg Oprozomib Tablet: Participants who were administered 180 mg oprozomib tablets.
- 210 mg Oprozomib Tablet: Participants who were administered 210 mg oprozomib tablets.
- 240 mg Oprozomib Tablet: Participants who were administered 240 mg oprozomib tablets.
- 270 mg Oprozomib Tablet: Participants who were administered 270 mg oprozomib tablets.
- 300 mg Oprozomib Tablet: Participants who were administered 300 mg oprozomib tablets.
- 150 mg Oprozomib ER Tablet: Participants who were administered 150 mg extended release oprozomib tablets.
- 300 mg Oprozomib ER Tablet: Participants who were administered 300 mg extended release oprozomib tablets.
- 330 mg Oprozomib ER Tablet: Participants who were administered 330 mg extended release oprozomib tablets.
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 9 | 9 | 4 | 6 | 5 | 3 | 19 | 6
hours | 1.0 [0.50 to 2.0] | 1.1 [0.50 to 6.0] | 1.0 [0.98 to 2.0] | 1.0 [0.50 to 2.0] | 2.0 [1.0 to 3.9] | 2.0 [1.1 to 4.0] | 1.0 [0.50 to 2.0] | 1.5 [0.47 to 4.0]

7. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Maximum Serum Concentration (Cmax) on Cycle 1, Day 1
Description: as for outcome 6
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 9 | 9 | 4 | 6 | 5 | 3 | 19 | 6
ng/mL | 633 (192.1) | 754 (91.7) | 841 (73.8) | 906 (69.3) | 881 (37.8) | 672 (54.5) | 785 (63.7) | 578 (80.1)

8. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Area Under the Curve at the Last Measurable Time Point (AUClast) on Cycle 1, Day 1
Description: The area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) was estimated using the linear trapezoidal method.
  PK samples obtained on the following schedule:
  Phase 1b Continuous Dosing, Cycles 1 and 2: Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 8 hours post-dose plus pre-dose on Day 2 Phase 1b Step-up Dosing, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2 Phase 2, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 9 | 9 | 4 | 6 | 5 | 3 | 19 | 6
hr*ng/mL | 1140 (197.4) | 1770 (104.7) | 2170 (51.8) | 1900 (68.9) | 2530 (63.4) | 1690 (16.1) | 1740 (70.3) | 1690 (70.8)

9. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Area Under the Curve From Time 0 to Time Infinity (AUCinf) on Cycle 1, Day 1
Description: The area under the plasma concentration-curve from time 0 to time infinity (AUCinf) was estimated using the linear trapezoidal method
  PK samples obtained on the following schedule:
  Phase 1b Continuous Dosing, Cycles 1 and 2: Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 8 hours post-dose plus pre-dose on Day 2 Phase 1b Step-up Dosing, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2 Phase 2, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 7 | 6 | 4 | 4 | 5 | 1 | 15 | 4
hr*ng/mL | 947 (229.7) | 1600 (127.2) | 2180 (51.6) | 1970 (88.8) | 2550 (63.5) | NA (NA) — calculation not performed for a single participant. | 1900 (77.7) | 2150 (27.6)

10. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Terminal Half-Life (t1/2,z) on Cycle 1, Day 1
Description: as for outcome 6
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 7 | 6 | 4 | 4 | 5 | 1 | 15 | 4
hr | 0.962 (40.6) | 0.573 (29.4) | 0.970 (79.2) | 0.850 (29.5) | 1.36 (80.1) | NA (NA) — calculation not performed for a single participant. | 0.710 (40.7) | 0.805 (40.1)

11. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Apparent Drug Clearance After Oral Administration (CL/F) on Cycle 1, Day 1
Description: The apparent drug clearance after oral administration (CL/F) was calculated as the dose divided by AUCinf.
  PK samples obtained on the following schedule:
  Phase 1b Continuous Dosing, Cycles 1 and 2: Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 8 hours post-dose plus pre-dose on Day 2 Phase 1b Step-up Dosing, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2 Phase 2, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 7 | 6 | 4 | 4 | 5 | 1 | 15 | 4
mL/hr | 190000 (229.7) | 131000 (127.2) | 110000 (51.6) | 137000 (88.8) | 118000 (63.5) | NA (NA) — calculation not performed for a single participant. | 157000 (77.7) | 153000 (27.6)

12. Secondary Outcome: Pharmacokinetic (PK) Parameter for Oprozomib, Tablet and ER Formulation: Apparent Volume of Distribution After Oral Administration (Vz/F) on Cycle 1, Day 1
Description: The apparent volume of distribution after oral administration (Vz/F) calculated as the dose divided by AUCinf times ƒz, where ƒz was the first-order terminal rate constant estimated via linear regression of the terminal log-linear phase.
  PK samples obtained on the following schedule:
  Phase 1b Continuous Dosing, Cycles 1 and 2: Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 8 hours post-dose plus pre-dose on Day 2 Phase 1b Step-up Dosing, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2 Phase 2, Day 1: pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, and 7 hours post-dose plus pre-dose on Day 2
Time Frame: Day 1
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | 180 mg Oprozomib Tablet | 210 mg Oprozomib Tablet | 240 mg Oprozomib Tablet | 270 mg Oprozomib Tablet | 300 mg Oprozomib Tablet | 150 mg Oprozomib ER Tablet | 300 mg Oprozomib ER Tablet | 330 mg Oprozomib ER Tablet
Number analyzed (Participants) | 7 | 6 | 4 | 4 | 5 | 1 | 15 | 4
mL | 264000 (235.6) | 108000 (106.7) | 154000 (79.5) | 168000 (138.9) | 231000 (54.7) | NA (NA) — calculation not performed for a single participant. | 161000 (69.0) | 178000 (44.3)

13. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Benefit Response As Assessed by Investigator During Phase 2
Description: The clinical benefit rate (CBR) was defined as Overall Response Rate (ORR) plus Minimal Response (MR) as defined by the European Group for Blood and Marrow Transplantation (EBMT) criteria.
Time Frame: Screening: Day 14 to Day -1; During study: Day 1 up to 13.16 months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
percentage of participants | 72.2 [46.5 to 90.3]

14. Secondary Outcome: Kaplan-Meier Estimates for Duration of Response (DOR) as Assessed by Investigator During Phase 2
Description: Duration of response was defined as the time from first evidence of partial response (PR) or better (i.e. best overall response) to confirmation of disease progression or death due to any cause. Durations were calculated for responders only. Medians and percentiles were estimated using the Kaplan-Meier method. 95% confidence intervals for medians and percentiles were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: Day 1 up to 13.16 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
months | NA [6.8 to NA] — not enough events to calculate

15. Secondary Outcome: Kaplan-Meier Estimates for Progression-free Survival (PFS) as Assessed by Investigator During Phase 2
Description: Progression-free survival (PFS) was defined as number of months between start of treatment and first evidence of documented disease progression or death (due to any cause), whichever occurs first. Disease progression was determined using IMWG-URC per investigator. The duration of PFS was right-censored for participants who met 1 of the following conditions:
  * 1) starting a new anticancer therapy before documentation of disease progression or death;
  * 2) death or disease progression immediately after more than 1 consecutively missed disease assessment visit or;
  * 3) alive without documentation of disease progression before the data cutoff date.
    95% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: Day 1 up to 14.1 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
months | 12.2 [3.5 to NA] — not enough events to calculate

16. Secondary Outcome: Kaplan-Meier Estimate for Time to Progression (TTP) as Assessed by Investigator During Phase 2
Description: Time to progression (TTP) was defined as the number of months between the start of treatment to the first documentation of disease progression. Disease progression was determined using IMWG-URC as assessed by the investigator. The same censoring rules, except for death, as in analysis of PFS were applied in the calculation of TTP.
  Participants who died prior to progressive disease were censored at the date of last evaluable response assessment.
Time Frame: Day 1 up to 14.1 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 300 mg 2/7 Schedule
Number analyzed (Participants) | 18
months | 12.2 [3.5 to NA] — not enough events to calculate

ADVERSE EVENTS:
Time Frame: All-cause Mortality - Death that occurred from the date of enrollment until the data cutoff of 30 July 2019. Treatment-emergent adverse events - Day 1 up to Week 282
Description: All-cause mortality is reported for all participants enrolled/randomized in the study.
  Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Phase 2 300 mg 2/7 Schedule: The Cohort Safety Review Committee (CSRC) determined this dose as the recommended phase 2 dose (RP2D). Oprozomib 300 mg once daily on Days 1, 2, 8, and 9 of a 14-day treatment cycle in combination with 20 mg dexamethasone once daily on Days 1, 2, 8, and 9 of a 14-day cycle. Treatment was administered in 14- day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason.
Arm/Group | Cohort 180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 5/14 Schedule (Phase 1b) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) | Cohort 210 mg 2/7 Schedule (Phase 1b) | Cohort 240 mg 2/7 Schedule (Phase 1b) | Cohort 270 mg 2/7 Schedule (Phase 1b) | Cohort 300 mg 2/7 Schedule (Phase 1b) | Cohort 330 mg 2/7 Schedule (Phase 1b) | Phase 2 300 mg 2/7 Schedule
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/7 | 0/3 | 0/4 | 1/4 | 0/6 | 0/8 | 0/6 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/9 | 2/7 | 2/3 | 2/4 | 1/4 | 1/6 | 3/8 | 0/6 | 9/18
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7 | 3/3 | 4/4 | 4/4 | 6/6 | 8/8 | 6/6 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 180 mg 5/14 Schedule (Phase 1b) (N=9) | Cohort 210 mg 5/14 Schedule (Phase 1b) (N=7) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) (N=3) | Cohort 210 mg 2/7 Schedule (Phase 1b) (N=4) | Cohort 240 mg 2/7 Schedule (Phase 1b) (N=4) | Cohort 270 mg 2/7 Schedule (Phase 1b) (N=6) | Cohort 300 mg 2/7 Schedule (Phase 1b) (N=8) | Cohort 330 mg 2/7 Schedule (Phase 1b) (N=6) | Phase 2 300 mg 2/7 Schedule (N=18)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 180 mg 5/14 Schedule (Phase 1b) (N=9) | Cohort 210 mg 5/14 Schedule (Phase 1b) (N=7) | Cohort 150/180 mg 5/14 Schedule (Phase 1b) (N=3) | Cohort 210 mg 2/7 Schedule (Phase 1b) (N=4) | Cohort 240 mg 2/7 Schedule (Phase 1b) (N=4) | Cohort 270 mg 2/7 Schedule (Phase 1b) (N=6) | Cohort 300 mg 2/7 Schedule (Phase 1b) (N=8) | Cohort 330 mg 2/7 Schedule (Phase 1b) (N=6) | Phase 2 300 mg 2/7 Schedule (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 1 | 1 | 0 | 5 | 3 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 1 | 2 | 3 | 2 | 4
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1 | 1 | 4 | 5 | 10
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 2 | 4 | 3 | 6 | 7 | 5 | 14
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 6
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 7 | 3 | 4 | 3 | 5 | 7 | 6 | 12
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5 | 3 | 4 | 3 | 2 | 2 | 5 | 8
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 8
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 3
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 6 | 4 | 2 | 2 | 2 | 4 | 7 | 6 | 7
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 5
Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 5
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 5 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 2 | 0 | 3 | 0 | 2 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 3 | 3 | 4
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 3 | 1 | 6
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 2 | 4
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic papillomatous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device implantation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT01832727/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT01832727/SAP_001.pdf